CLINICAL TRIAL: NCT02786329
Title: The Influence of Anesthesia on Postoperative Outcome and Complications in Colorectal Cancer Patients
Brief Title: Anesthesia and Postoperative Outcome in Colorectal Cancer Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Collaborators: Prof. Dr. I. Chiricuta Institute of Oncology (Other)
Responsible Party: Principal Investigator, Prof.Dr.Daniela Ionescu, Professor, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 53/14.03.2016
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; TIVA; sevoflurane; lidocaine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TIVA + lidocaine (Active Comparator): TIVA-L. Patients allocated to receive TIVA (propofol-fentanyl) with lidocaine infusion.
  Interventions: TIVA+lidocaine
  Interventions: Drug: TIVA+lidocaine
- TIVA+placebo (Placebo Comparator): TIVA-P. Patients allocated to receive TIVA without lidocaine (placebo). Intervention: TIVA+placebo (saline infusion)
  Interventions: Drug: TIVA+placebo
- Sevoflurane+placebo (Placebo Comparator): Sevo-P. Patients allocated to receive Sevoflurane anesthesia without lidocaine infusion (placebo).
  Intervention: sevoflurane anesthesia +placebo (saline infusion)
  Interventions: Drug: Sevoflurane+placebo
- Sevoflurane+lidocaine (Active Comparator): Sevo-L. Patients allocated to receive sevoflurane anesthesia with lidocaine infusion for the first 48 h postoperatively.
  Intervention: sevoflurane anesthesia+ lidocaine infusion
  Interventions: Drug: Sevoflurane+lidocaine

INTERVENTIONS:
Drug: TIVA+lidocaine — Patients will be subjected to total intravenous anesthesia with propofol-fentanyl+i.v. lidocaine infusion for the first 48 h postoperatively
  Other Names: TIVA-L
  Arms: TIVA + lidocaine
Drug: Sevoflurane+lidocaine — Patients will be subjected to anesthesia with sevoflurane- fentanyl + lidocaine infusion for the first 48 h postoperatively.
  Other Names: Sevo-L
  Arms: Sevoflurane+lidocaine
Drug: TIVA+placebo — Patients will be subjected to TIVA with propofol-fentanyl + saline infusion for the first 48 h postoperatively
  Other Names: TIVA-P
  Arms: TIVA+placebo
Drug: Sevoflurane+placebo — Patients will be subjected to anesthesia with sevoflurane-fentanyl + saline infusion for the first 48 h postoperatively
  Other Names: Sevo-P
  Arms: Sevoflurane+placebo

SUMMARY:
Study aims to compare the influence of TIVA and sevoflurane anesthesia with or without lidocaine on postoperative short and long term outcome in patients with colorectal cancer undergoing surgery.

As short term endpoints postoperative pain and opioid consumption, resumption of bowel function, PONV, LOS will be registered.

Long term outcome parameters include: the incidence of chronic pain, 1 and 5 years cancer recurrences incidence and mortality.

DETAILED DESCRIPTION:
Main goals

1. Comparative evaluation of the incidence of recurrences after TIVA vs sevoflurane anesthesia
2. Evaluation of the effect of lidocaine infusion associated with TIVA/sevoflurane on the incidence of chronic pain and of cancer recurrences and survival.

Secondary objectives

1. Evaluation of the influence of lidocaine on postoperative outcome in patients with colorectal cancer
2. Evaluation of the influence of lidocaine on postoperative inflammatory response
3. Evaluation of the influence of lidocaine on the incidence and severity of postoperative pain and outcome in patients with colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery

Exclusion Criteria:

* • persistent chronic pain

  * chronic medication that may interfere with pain: antiepileptics, NSAID, corticoids
  * Contraindications for any of the study medications
  * Significant psychiatric disorders (Axa I) (major depression, bipolar disorders, schizophrenia, etc.)
  * Significant hepatic (ALAT and/or ASAT > 2 normal values) or renal (plasma creatinine > 2 mg/dl) disorders
  * Convulsive disorders requiring medication during the last 2 years
  * Planned regional analgesia/anesthesia (spinal or epidural)
  * Corticoid dependent asthma
  * Autoimmune disorders
  * Anti-arrhythmic medication (verapamil, propafenone, amiodarone) that may interfere with lidocaine's anti-arrhythmic effects
  * Refusal for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Survival after TIVA vs sevoflurane anesthesia in patients operated for colorectal cancer | 5 years
  Survival at 5 years will be recorded
Incidence of recurrences: | 5 years
  The incidence of recurrences will be registered annually and reported from the first year to 5 years respectively in all 4 groups of patients.

SECONDARY OUTCOMES:
Morphine consumption during the first 24 postoperative hours | 0- 24 h
  Total morphine consumption during the first 24h after surgery will be recorded
Severity of postoperative pain - verbal response pain (VRPS) score 1-10, (1=no pain, 10=worst pain) in recovery room and during the first 48 hrs postoperatively. Target verbal response pain score ≤3 | 0- 48 h
  The severity of postoperative pain will be recorded along with morphine consumption.Pain intensity will be followed during the first 48 h postoperatively.
Resumption of bowel function | 0-72 h
  Time to first flatus will be registered and compared between groups.
Length of hospital stay | 0-10 days
  LOS will be registered and compared between study groups.
Postoperative chronic pain | 1 year
  Chronic pain at 6 month and 1 year respectively will be assessed with McGill questionnaire by telephone interview.
  Scores range from 0 (no pain) to 78 (severe pain), patients with high scores need to seek medical advice
Postoperative imflamation | Day 1
  Evaluation of the influence of lidocaine on 24-hour postoperative inflammatory response; All patients will have leukocytes count and c protein reactive (PCR) so an analysis can be made.
Rate of postoperative complications after intravenous lidocaine infusion versus placebo | 0-30 days
  Monitoring the incidence of some common perioperative complications: pulmonary embolism, pulmonary edema, acute kidney injury, anastomosis leak, myocardial infarction, stroke, pneumonia
Rate of postoperative complications after TIVA versus inhalation anaesthesia | 0-30 days
  Monitoring the incidence of some common perioperative complications: pulmonary embolism, pulmonary edema, acute kidney injury, anastomosis leak, myocardial infarction, stroke, pneumonia

OTHER OUTCOMES:
Rate of local anaesthetics systemic toxicity incidence | 0-48 hours
  An investigator will note any signs of local anaesthetics systemic toxicity at the bed site of patient

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, Prof, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca; Alexandru Alexa, Assist Prof, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca
Locations (2):
- Romania (2):
  - Clinica ATI, str Croitorilor nr 19-21, Cluj-Napoca, Cluj
  - Institutul Oncologic Prof Dr Ion Chiricuta, Cluj-Napoca, Cluj

IPD SHARING:
Plan to Share IPD: Yes
Regular meeting for sharing data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be shared between cooperation institutions every 3 month and whenever necessary.
Access Criteria: Access criteria are: active involvement into the study, the need to register data into the common database.
  The need to report data into the PhD thesis is also an access criteria.

REFERENCES:
- [Background] Fodale V, D'Arrigo MG, Triolo S, Mondello S, La Torre D. Anesthetic techniques and cancer recurrence after surgery. ScientificWorldJournal. 2014 Feb 6;2014:328513. doi: 10.1155/2014/328513. eCollection 2014. PMID 24683330
- [Background] Heaney A, Buggy DJ. Can anaesthetic and analgesic techniques affect cancer recurrence or metastasis? Br J Anaesth. 2012 Dec;109 Suppl 1:i17-i28. doi: 10.1093/bja/aes421. PMID 23242747
- [Background] Mao L, Lin S, Lin J. The effects of anesthetics on tumor progression. Int J Physiol Pathophysiol Pharmacol. 2013;5(1):1-10. Epub 2013 Mar 8. PMID 23525301
- [Background] Cakmakkaya OS, Kolodzie K, Apfel CC, Pace NL. Anaesthetic techniques for risk of malignant tumour recurrence. Cochrane Database Syst Rev. 2014 Nov 7;2014(11):CD008877. doi: 10.1002/14651858.CD008877.pub2. PMID 25379840
- [Background] Cassinello F, Prieto I, del Olmo M, Rivas S, Strichartz GR. Cancer surgery: how may anesthesia influence outcome? J Clin Anesth. 2015 May;27(3):262-72. doi: 10.1016/j.jclinane.2015.02.007. Epub 2015 Mar 11. PMID 25769963
- [Background] Divatia JV, Ambulkar R. Anesthesia and cancer recurrence: What is the evidence? J Anaesthesiol Clin Pharmacol. 2014 Apr;30(2):147-50. doi: 10.4103/0970-9185.129990. No abstract available. PMID 24803747
- [Result] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Result] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Derived] Alexa AL, Tat TF, Ionescu D. The influence of TIVA or inhalation anesthesia with or without intravenous lidocaine on postoperative outcome in colorectal cancer surgery: a study protocol for a prospective clinical study. Trials. 2022 Mar 18;23(1):219. doi: 10.1186/s13063-022-06157-4. PMID 35303929